CLINICAL TRIAL: NCT05200546
Title: Improving Carbapenemase-Producing Organism (CPO) and Vancomycin-Resistant Enterococcus (VRE) Management With BD Solutions
Brief Title: Carbapenemase-Producing Organism and Vancomycin-Resistant Enterococcus Management
Acronym: CPO-VRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0370; 2021-A02468-33 (Other: ID RCB)
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Multidrug-resistant Bacteria Screening
Keywords: mutlidrug resistant bacteria; carbapenemase-producing enterobacteria; vancomycin-resistant enterococci; molecular assays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group "before": 1st period of 6 months during which only the current detection technique will be used.
- group "after": - 2nd period of 6 months after implementation of the PCR solution (CPO and VRE) of the BD company in parallel with the usual screening technique
  Interventions: Diagnostic Test: molecular assays to screen for eXDR

INTERVENTIONS:
Diagnostic Test: molecular assays to screen for eXDR — VRE detection will be performed using "VIASURE Vancomycin resistance Real Time PCR Detection Kit".
  BD MAX Check-Points CPO will be used to detect carbapenemase-producing organisms.
  Groups: group "after"

SUMMARY:
Emergence of vancomycin-resistant enterococci (VRE) and carbapenemase-producing enterobacteria (CPE) is nowadays a major public health concern worldwide. VRE and CPE are referred to as Emerging eXtensively Drug Resistant bacteria (eXDR).

A better, faster and more accurate identification of VRE and CPE would allow faster appropriate therapy for patients and/or infection control strategies. Faster appropriate therapy could improve mortality rates, length of stay, and other patient outcomes as well as hospital costs. BD offers a variety of products, services and solutions designed to increase efficiency, streamline processes, and deliver high quality and consistent results with improved turnaround time.

The primary objective of this study will be to measure the impact of the BD CPO and VRE PCRs on the turnaround time for eXDR positive detection.

Study will collect criteria and compared several outcomes before and after the implementation of the BD solutions for the detection of eXDR.

This is a non-interventional research with a before/after design.

The study therefore consists of two periods:

* 1st period of 6 months during which only the current detection technique will be used.
* 2nd period of 6 months after implementation of the PCR solution (CPO and VRE) of the BD company in parallel with the usual screening technique.

Advantages of using molecular assays to screen for eXDR include labor savings, faster turnaround time, and higher sensitivity than culture-based methods.

In trying to reduce testing time, investigators should have better control of the eXDR transmission. this should reduce patient-to-patient transmissions. The number of contact patient in case of one positive screening should decrease. The number of days where patients are unnecessary placed in preemptive isolation should also decrease.

Moreover, PCR will be use in first intention and only positive samples in PCR will be cultivated; For the laboratory, technician time saving is expected given the simplicity of the PCRs. Plate readings at 24 and 48h will be limited to a few samples. Investigators also expect a significant gain in financial terms for hospital by performing a medico-economic analysis. According to the shorter time for getting results using BD solution in diagnosing patients at risk, investigators then assume that a shorter time in making clinical decision will be a normal consequence, and will imply a better relevant organization of care with lower real costs.

DETAILED DESCRIPTION:
Carbapenemases, with versatile hydrolytic capacity against β-lactams, are now an important cause of resistance of Gram-negative bacteria. Furthermore, they are often resistant to a wide-range of antimicrobial agents The genes encoding for the acquired carbapenemases are associated with a high potential for dissemination. In addition, infections due to Gram-negative bacteria with acquired carbapenemase production would lead to high clinical mortality rates. These organisms often render standard empiric therapy ineffective. In fact, Zilberberg et al. demonstrated a higher rate of inappropriate empiric therapy leading to increased length of stay, mortality risk and hospital costs for carbapenem resistant organisms vs susceptible organisms.

The control of the VRE emergence became a priority to tackle the antibiotic resistance, fearing a transfer of the resistance to the methicillin-resistant Staphylococcus aureus (MRSA). VRE outbreaks were reported in CHUGA. Because of the high transmission potential, those VRE outbreaks had a substantial impact on the healthcare activity.

Hypothesis: a better, faster and more accurate identification of VRE and CPE would allow faster appropriate therapy for patients and/or infection control strategies. Faster appropriate therapy could improve mortality rates, length of stay, and other patient outcomes as well as hospital costs.

The primary objective of this study will be to measure the impact of the BD CPO and VRE PCRs on the turnaround time for eXDR positive detection.

A before and after study design will be used. Investigators will compare the average turnaround time before and after the implementation of BD solutions.

Turnaround time is defined as time from sample collection to result delivered to the clinician and/or infection control team.

Result is defined as the detection of the major carbapenemase genes, including blaKPC, blaOXA-48, blaVIM and blaNDM genes or the detection of vanA gene associated to E. faecium identification from fecal swabs.

ELIGIBILITY:
Inclusion Criteria:

Anybody coming in the CHUGA with at least one criteria of eXDR screening:

* Hospitalized patients at least two times within the previous year
* Patient transferred from another hospital
* Patient transferred from nursing home
* Patient with a history of hospitalization abroad (foreign countries) within the previous year
* Contact patient = patient exposed to an eXDR bacteria carrier
* eXDR carrier

Exclusion Criteria:

* Refusal to participate to the study. Opposition of the patients to the use of their personal data.
* Refusal of rectal swab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anybody coming in the CHUGA with at least one criteria of eXDR screening
Sampling Method: Non-Probability Sample
Enrollment: 3921 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
impact of the BD CPO and VRE PCRs on the turnaround time for eXDR positive detection | 12 months
  Compare the average turnaround time before and after the implementation of BD solutions.
  Turnaround time is defined as time from sample collection to result delivered to the clinician and/or infection control team.
  Result is defined as the detection of the major carbapenemase genes, including blaKPC, blaOXA-48, blaVIM and blaNDM genes or the detection of vanA gene associated to E. faecium identification from fecal swabs.

SECONDARY OUTCOMES:
impact of the BD CPE and VRE PCR on the number of rectal screening performed by the laboratory | 12 months
  Comparison before and after the implementation of BD solutions of the average number of rectal screening
turnaround time of removal of isolation measure | 12 months
  In case of negative results, the turnaround time of removal of isolation measure for patients with a history of hospitalization abroad within the previous year will be determined.
number of patients in contact with eXDR patients | 12 months
  In case of positive results, the average number of patients in contact with the eXDR carrier will be determined.
number of eXDR secondary cases | 12 months
  The average number of secondary eXDR cases will be compared before and after the implementation of BD solutions.
number of day where the transfers and admissions are blocked for a medical unit | 12 months
  The average number of day where the transfers and admissions are blocked for a medical unit will be compared before and after the implementation of BD solutions.
real cost of tests solutions | 12 months
  The real cost of tests solutions, regarding to the amount of reimbursement by health insurance will be estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine BOISSET, Principal Investigator — UGA, CHUGA
Locations (1):
- Grenoble_Alpes UniversityHospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zilberberg MD, Shorr AF, Micek ST, Vazquez-Guillamet C, Kollef MH. Multi-drug resistance, inappropriate initial antibiotic therapy and mortality in Gram-negative severe sepsis and septic shock: a retrospective cohort study. Crit Care. 2014 Nov 21;18(6):596. doi: 10.1186/s13054-014-0596-8. PMID 25412897
- [Background] Bilavsky E, Schwaber MJ, Carmeli Y. How to stem the tide of carbapenemase-producing enterobacteriaceae?: proactive versus reactive strategies. Curr Opin Infect Dis. 2010 Aug;23(4):327-31. doi: 10.1097/QCO.0b013e32833b3571. PMID 20581673
- [Background] Zilberberg MD, Nathanson BH, Sulham K, Fan W, Shorr AF. 30-day readmission, antibiotics costs and costs of delay to adequate treatment of Enterobacteriaceae UTI, pneumonia, and sepsis: a retrospective cohort study. Antimicrob Resist Infect Control. 2017 Dec 6;6:124. doi: 10.1186/s13756-017-0286-9. eCollection 2017. PMID 29225798
- [Background] Lepelletier D, Berthelot P, Lucet JC, Fournier S, Jarlier V, Grandbastien B; National Working Group. French recommendations for the prevention of 'emerging extensively drug-resistant bacteria' (eXDR) cross-transmission. J Hosp Infect. 2015 Jul;90(3):186-95. doi: 10.1016/j.jhin.2015.04.002. Epub 2015 Apr 24. PMID 25986165
- [Background] Mak A, Miller MA, Chong G, Monczak Y. Comparison of PCR and culture for screening of vancomycin-resistant Enterococci: highly disparate results for vanA and vanB. J Clin Microbiol. 2009 Dec;47(12):4136-7. doi: 10.1128/JCM.01547-09. Epub 2009 Oct 21. PMID 19846635
- [Background] Holzknecht BJ, Hansen DS, Nielsen L, Kailow A, Jarlov JO. Screening for vancomycin-resistant enterococci with Xpert(R) vanA/vanB: diagnostic accuracy and impact on infection control decision making. New Microbes New Infect. 2017 Jan 12;16:54-59. doi: 10.1016/j.nmni.2016.12.020. eCollection 2017 Mar. PMID 28203378